CLINICAL TRIAL: NCT05711771
Title: Medication Therapy Management (MTM) for a Medicaid Managed Care Population Within Patient-Centered Medical Homes
Status: Withdrawn | Type: Observational
Sponsor: Ohio State University (Other)
Responsible Party: Principal Investigator, Kelli Barnes, Assistant Professor - Clinical, Ohio State University
Other Study IDs: #2014H0382
Record Dates: First submitted 2015-03-18; First posted 2023-02-03 (Actual); Last update posted 2023-02-03 (Actual); Status verified 2023-01

CONDITIONS: Medication Therapy Management; Estimated Cost Avoidance; MTM; Medication Management
MeSH Terms: interventions — Medication Therapy Management

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Behavioral: medication therapy management — Patients receive medication therapy management within the primary care office

SUMMARY:
The primary objective of this project is to determine the estimated cost avoidance (ECA) resulting from medication therapy management (MTM) interventions in a patient-centered medical home (PCMH). The secondary objective of this study is to quantify the number and types of MTM interventions recommended by pharmacists and accepted by physicians within a PCMH.

DETAILED DESCRIPTION:
CareSource™, the largest Medicaid managed care provider in Ohio, pays for pharmacist-provided MTM using the OutcomesMTM™ platform for claims submissions. In May of 2013, pharmacists at three PCMHs affiliated with a large academic medical center began providing MTM to patients with CareSourceTM through the OutcomesMTMTM platform. A retrospective chart review of the OutcomesMTM™ platform was performed for all patients who received MTM services between May 2013 and October 2014. The number and type of MTM interventions was tracked. For each intervention, the ECA level submitted to and accepted by the third party reviewer was collected. The ECA will be calculated using the cost associated to the CareSource™ managed care provider for each ECA level.

ELIGIBILITY:
Inclusion Criteria:

* Patient of a primary care doctor within The Ohio State University Division of General Internal Medicine
* CareSource™ Medicaid managed care as the insurance provider

Exclusion Criteria:

* n/a

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients of the CareSource™ Medicaid managed care population who have a primary care physician within the patient-centered medical homes of The Ohio State University Division of General Internal Medicine
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2015-02; Primary Completion 2015-12 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
Estimated cost avoidance | 1.5 years of data collected retrospectively

SECONDARY OUTCOMES:
Number of medication therapy management claims made | 1.5 years of data collected retrospectively
Types of medication therapy management claims made | 1.5 years of data collected retrospectively